CLINICAL TRIAL: NCT06976710
Title: Virtual Multimodal Hub for Patients Undergoing Colorectal Cancer Surgery - PRIORITY-CONNECT 2 Randomised Type I Hybrid Effectiveness-Implementation Trial
Brief Title: PRIORITY-CONNECT 2 Trial
Acronym: PC2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Surgical Outcomes Research Centre (SOuRCe) (Network)
Collaborators: The University of Sydney, Sydney, Australia (Unknown); Medical Research Future Fund (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: X23-0399 Phase 2
Record Dates: First submitted 2025-04-13; First posted 2025-05-16 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Cancer; Colorectal Neoplasms
Keywords: Prehabilitation; Colorectal Cancer; Surgery; Surgical Outcomes; Randomised Controlled Trial; Virtual Rehabilitation; Virtual Prehabilitation; Multidisciplinary; Virtual Care; Rehabilitation
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Preoperative Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The randomisation sequence will be prepared a priori using a central secure randomisation service (1:1 allocation ratio in random permuted blocks of sizes 4 or 2 stratified by hospital, to ensure balance in treatment assignment within hospital) to ensure concealment of treatment allocation and blinding of surgeon, all trial personnel, health economist and statistician. Due to the nature of the intervention, it is not possible to blind the clinicians delivering the intervention (virtual multimodal hub); however, the investigators will ensure that all patients' interactions are standardised according to standard operating procedures (SOPs).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Multimodal Hub and usual care (Intervention Group) (Experimental): The intervention is a multicomponent virtual hub which encompasses medical, social, psychological and functional assessment(s) and intervention(s). Following a comprehensive holistic assessment, clinicians will tailor the intervention subject to individual's presentation and needs. This may include evidence-based exercise, nutritional, psychological and nursing interventions, and /or group-delivered peer support, in addition to usual care. Adjustments and progression will be made in each session according to an individual's response. All interventions will be conducted before and after surgery.
  Standardised assessment tools will guide the frequency, intensity, duration, type, volume, and progression of the multimodal interventions, with the potential for the intervention(s) to be stepped-up or stepped-down based on individual patient needs
  Interventions: Behavioral: Preoperative Exercise; Behavioral: Postoperative Exercise; Dietary Supplement: Preoperative Nutrition; Dietary Supplement: Postoperative Nutrition; Behavioral: Preoperative Psychology; Behavioral: Postoperative Psychology; Other: Preoperative Nursing; Other: Postoperative Nursing; Behavioral: Preoperative Peer Support Group; Behavioral: Postoperative Peer Support Group; Other: Usual Care
- Usual care alone (Control Group) (Active Comparator): Participants allocated to the control group will only receive usual care according to their health care team, which may consist of advice on smoking cessation, reduction of alcohol intake, nutritional counselling, and medical optimisation in the preoperative anaesthetic clinic visits. Participants will be asked to maintain their normal daily activities. No attempt will be made to alter the routine care pathway. The use of any additional service will be recorded to inform the comprehensive cost analysis (linked to PBS and MBS data).
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Preoperative Exercise — Aerobic, Endurance, Respiratory, Muscle Strength, Education
  Arms: Virtual Multimodal Hub and usual care (Intervention Group)
Behavioral: Postoperative Exercise — Aerobic, Endurance, Respiratory, Muscle Strength, Education
  Arms: Virtual Multimodal Hub and usual care (Intervention Group)
Dietary Supplement: Preoperative Nutrition — Malnutrition screening, Weight monitoring, Symptom management, Dietetic counselling, Nutrition support
  Arms: Virtual Multimodal Hub and usual care (Intervention Group)
Dietary Supplement: Postoperative Nutrition — Malnutrition screening, Weight monitoring, Symptom management, Dietetic counselling, Nutrition support
  Arms: Virtual Multimodal Hub and usual care (Intervention Group)
Behavioral: Preoperative Psychology — CBT skills, Skills training, Emotional validation, Behavioural activation, Psycho-education
  Arms: Virtual Multimodal Hub and usual care (Intervention Group)
Behavioral: Postoperative Psychology — CBT skills, Skills training, Emotional validation, Behavioural activation, Psycho-education
  Arms: Virtual Multimodal Hub and usual care (Intervention Group)
Other: Preoperative Nursing — Risk management, Managing pain, Wound care, Bowel function, Surgical education
  Arms: Virtual Multimodal Hub and usual care (Intervention Group)
Other: Postoperative Nursing — Risk management, Managing pain, Wound care, Bowel function/Stoma management, Education
  Arms: Virtual Multimodal Hub and usual care (Intervention Group)
Behavioral: Preoperative Peer Support Group — Fortnightly sessions moderated by a social worker including patients and carers:
  Safe space, Share experiences/ideas, Support, Education
  Arms: Virtual Multimodal Hub and usual care (Intervention Group)
Behavioral: Postoperative Peer Support Group — Fortnightly sessions moderated by a social worker including patients and carers:
  Safe space, Share experiences/ideas, Support, Education
  Arms: Virtual Multimodal Hub and usual care (Intervention Group)
Other: Usual Care — All participants will receive usual care according to their health care team, which may consist of advice on smoking cessation, reduction of alcohol intake, nutritional counselling, and medical optimisation in the preoperative anaesthetic clinic visits.

SUMMARY:
Objectives:

The primary aim of this project is to establish the effectiveness of an individualised stepped, multidisciplinary intervention, including education and peer support group, delivered via a virtual multimodal (p)rehabilitation hub, in reducing postoperative complications within 30-days following colorectal cancer surgery, compared to usual care alone.

The secondary aims will be to obtain data on the likely difference in key outcomes including:

(i) Quality of life (EORTC QLQ-C30 and QLQ-CR29) (ii) Number of days at home within 30, 90 and 365 days after surgery (DAH-30, 90, 365) (iii) Quality of recovery (QoR-15) (iv) Cost-effectiveness (v) Implementation metrics (RE-AIM)

Our hypothesis is that the PRIORITY-CONNECT 2 intervention will be more effective in reducing postoperative complications and more cost-effective than usual care.

Study design:

Pragmatic Randomised Type I Hybrid Effectiveness-Implementation Trial.

Planned sample size:

To achieve the primary aim, 564 participants will provide 90% power to detect a 15% difference in 30-day postoperative complication rates between the intervention and control groups. The sample size calculation accounts for up to 10% loss to follow-up, 5% non-compliance and a two-side alpha of 0.05.

Selection criteria:

A sample of 564 participants undergoing colorectal cancer surgery including open, laparoscopic or robotic-assisted surgery (mostly, anterior resection, sigmoid colectomy, hemicolectomy, total proctocolectomy, subtotal colectomy, total colectomy) at sites throughout Australia will be included. These are common colorectal cancer surgeries performed at the participating centres. All the surgeons involved in this study have clinical appointments in their respective hospitals.

Inclusion: Adults aged ≥18 years undergoing elective major surgery for colon or rectal cancer with curative intent; and consulting a colorectal surgeon at least 1 week prior to scheduled surgery.

Exclusion: Patients undergoing Pelvic Exenteration (PE), Cytoreductive Surgery (CRS) with or without HIPEC, or concurrent surgery for metastatic disease; or cognitive impairment such that they are unable to provide informed consent.

Study Procedure:

Participant's treating team will screen and provide an information sheet about the trial to consecutive patients. Interested patients will be contacted by a study researcher to discuss the trial further, answer any questions, confirm eligibility against the inclusion and exclusion criteria, and consent patients. Consenting patients will undergo baseline assessment and be randomised to a virtual multimodal hub (Intervention group) or usual care alone (Control group). The intervention will include the delivery of usual care and evidence-based exercise, nutritional, psychological and nursing interventions, and / or group-delivered peer support. All interventions will be conducted before and after surgery.

Duration of the Study:

Approximately 60 months.

Funding:

Medical Research Future Fund (MRFF) 2023 Early and Mid-Career Researchers (Application ID: 2031563).

Sponsor:

The University of Sydney.

DETAILED DESCRIPTION:
Further details on the study procedures:

Patients will be identified by their treating team (including but not limited to colorectal surgeon, allied health, research and nursing staff). The treating team will screen and provide the information sheet about the trial to consecutive patients. Interested patients will be contacted by a study researcher to discuss the trial further, answer any questions, confirm eligibility against the inclusion and exclusion criteria, and consent patients. Consenting patients will undergo baseline assessment and be randomised to a virtual multimodal hub (Intervention group) or usual care alone (Control group). Patients will undergo an immediate second randomisation to determine their virtual hub assignment (Royal Prince Alfred Hospital Hub or The Peter MacCallum Cancer Centre Hub).

The participants randomised into the intervention group will then be contacted by a range of allied health workers, depending on their individual needs. These may include a physiotherapist, dietitian, psychologist, nurse and/ or a social worker. The intervention will provide the participants support as they navigate the health system. These health workers will communicate with them via the virtual hub for sessions to provide support before surgery and help with their recovery. Participant's individual needs will determine the frequency, intensity, time, type, volume, and progression of these sessions. This intervention may last for up to 12 months after their surgery, but they will be discharged from the intervention once they have reached their treatment goals. If participants do not have access to a smart device and/or internet, the investigators can provide them with a tablet with internet connectivity to engage in virtual delivery of sessions.

Data and safety monitoring:

An independent Data and Safety Monitoring Board (DSMB), will be monitored by a multidisciplinary panel (including statistician(s)). This panel will assess for adverse events and adherence to the protocol at regular intervals to ensure the safety of participants. The frequency of DSMB meetings and the stopping rules for the study will be defined a priori in a charter, in consultation with the DSMB members and study investigators. This will include after commencing participant recruitment and once one fourth of participants have been recruited.

ProCoMida:

The PRO CoMiDa form is a data management tool, designed to provide standardised documentation of the completion, or reasons for non-completion, of patient reported outcomes assessments by patients in a clinical trial. Such documentation is crucial for quality assurance since missing data is the greatest threat to the integrity and interpretability of patient reported outcomes data. The PRO CoMiDa form must be completed at each scheduled patient reported outcomes assessment.

GCP Certificates:

The trial will conform to all relevant ICH GCP guidelines and regulations. Annual audits will be conducted by research officers to ensure that all study staff maintain current GCP certification.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥18 years undergoing elective major surgery for colon or rectal cancer with curative intent
* Consulting with a colorectal cancer surgeon at least 1 week prior to scheduled surgery

Exclusion Criteria:

* Patients undergoing Pelvic Exenteration (PE), Cytoreductive Surgery (CRS) with or without HIPEC, or concurrent surgery for metastatic disease
* Cognitive impairment such that they are unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 564 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2028-07-30 (Estimated); Study Completion 2028-07-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants developing postoperative complications within 30 days after surgery. | First 30-days after surgery
  The primary outcome will be the proportion of participants developing postoperative complications within 30 days after surgery, defined as any deviation from the normal postoperative course and classified according to the Clavien-Dindo classification. The risk of developing complications following colorectal cancer surgery is highest in the first 30-days after surgery; this is a critical determinant of recovery, long-term outcomes, and colorectal cancer treatment costs.

SECONDARY OUTCOMES:
Quality of Life Outcome (EORTC QLQ-C30 and QLQ-CR29) | Measured at baseline, 1-2 day(s) before surgery, perioperative (within 1 day of hospital discharge), 1, 3, 6 and 12 months post index surgery.
  The European Organization for the Research and Treatment of Cancer (EORTC) Quality of Life Questionnaires (QLQ) are validated, cancer-specific tools commonly used to assess quality of life in colorectal cancer patients. The QLQ-C30 includes 30 items assessing five functional domains, nine symptom scales, financial impact and overall quality of life. The QLQ-CR29 is a 29-item tool to evaluate symptoms (gastrointestinal, urinary, pain and others) and functional areas (sexual, body image and others) that are associated with colorectal cancer and its treatments. Both tools use scales ranging from 0 to 100. Higher scores on functional and global health scales reflect better functioning or quality of life, whereas higher scores on symptom scales indicate greater symptom burden or problems.
Quality of Recovery (QoR-15) | Measured at baseline, 1-2 day(s) before surgery, perioperative (within 1 day of hospital discharge), 1, 3, 6 and 12 months post index surgery.
  The QoR-15 is a validated tool designed to assess the quality of recovery after surgery. It consists of 15 items rated on an 11-point numerical rating scale ranging from 0 to 10. The overall QoR-15 score is calculated by summing all individual item scores, resulting in a total score ranging from 0 to 150, where higher scores indicate a better quality of recovery. Recovery will be defined as return to baseline values or better in each of the questions or assessments.
Number of days at home within 30, 90 and 365 days of surgery (DAH-30, 90, 365) | Days at home within 30, 90 and 365 days of index surgery
  Validated (Australian-population) patient-centred outcome metrics that integrates length of hospital stay, discharge destination (other than home), hospital readmission and early death. The number of days at home is reduced by, for example, complications elongating acute hospital bed stay, discharge to a care facility, re-admission, and death. This is quantified as the days alive and at home during the 30 days after surgery. Days at home is calculated using mortality and hospitalisation data from the date of the index surgery (= Day 0).
Resource use (costs) | Measured at baseline, 1, 3, 6 and 12 months post index surgery.
  Patient and health system resource use, including the cost of the virtual multimodal hub interventions, hospitalisations, will be collected (surveys) from randomisation (1-6 weeks prior to surgery) to 12 months post index surgery.
Implementation metrics: (RE-AIM) | Through study completion, an average of 12 months
  The framework is used to plan, evaluate and assess the impact of a variety of health care and prevention programs. Elements assessed: Reach: Proportion of eligible patients recruited into the study, alongside the baseline characteristics (referral pathways, age, postcode, marital, work status, and cultural and linguistic diversity) of all potential participants. Effectiveness: Clinical outcomes, healthcare utilisation, and participant satisfaction (measured both quantitatively and qualitatively). Adoption: Referral rates, enablers and barriers (collected post intervention from patients, carers, surgeons, clinical and administrative staff). Implementation: Centre level - implementation process (patients, carers, and clinical staff interviews and direct observation), concordance with intervention protocol. Maintenance: referral rates and stakeholder interviews to identify refinements and infrastructure needed to maintain and scale intervention beyond the project period.

OTHER OUTCOMES:
Pain (NPRS) | Measured at baseline, 1-2 day(s) before surgery, perioperative (within 1 day of hospital discharge), 1, 3, 6 and 12 months post index surgery.
  The Numeric Pain Rating Scale (NPRS) is a widely used tool for assessing pain intensity in individuals. It is a segmented numeric scale where respondents select a whole number (0-10) that best reflects their pain intensity. The scale ranges from 0, indicating "no pain," to 10, representing "the worst pain imaginable." This method allows for a straightforward and quantifiable measure of pain, facilitating communication between patients and healthcare providers.
Exercise capacity (30sSTS) | Measured at baseline, 1-2 day(s) before surgery, perioperative (within 1 day of hospital discharge), 1, 3, 6 and 12 months post index surgery.
  30 seconds Sit-to-Stand Test (30sSTS) is a reliable and valid tool in evaluating functional exercise capacity in patients.The 30sSTS the performance of as many sit-to-stand actions as possible in 30 seconds without upper limb involvement.
Self-reported physical activity (IPAQ-SF) | Measured at baseline, 1-2 day(s) before surgery, perioperative (within 1 day of hospital discharge), 1, 3, 6 and 12 months post index surgery.
  International Physical Activity Questionnaire short form (IPAQ-SF) measures the types of intensity of physical activity and sitting time that people do as part of their daily lives. The questionnaire asks participants to report any physical activity (performed for at least 10 minutes) during the last seven days reported as hours per day, minutes per day, and days per week. This aims to be an estimate of total physical activity. IPAQ-SF has demonstrated high reliability and validity.
Nutritional Status (PG-SGA SF) | Measured at baseline, 1-2 day(s) before surgery, perioperative (within 1 day of hospital discharge), 1, 3, 6 and 12 months post index surgery.
  Patient-Generated Subjective Global Assessment Short Form (PG-SGA SF) includes four patient-generated historical components (Weight History, Food Intake, Symptoms and Activities and Function).
Anxiety (GAD-7) | Measured at baseline, 1-2 day(s) before surgery, perioperative (within 1 day of hospital discharge), 1, 3, 6 and 12 months post index surgery.
  General Anxiety Disorder-7 (GAD-7) is a self-administered patient questionnaire used as a screening tool and severity measure for generalised anxiety disorder (GAD). Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively.
Depression (PHQ-9) | Measured at baseline, 1-2 day(s) before surgery, perioperative (within 1 day of hospital discharge), 1, 3, 6 and 12 months post index surgery.
  Patient Health Questionnaire-9 (PHQ-9) is a self-administered version of the PRIME-MD diagnostic instrument for common mental disorders.The PHQ-9 is the depression module, which scores each of the nine DSM-IV criteria as "0" (not at all) to "3" (nearly every day). PHQ-9 is used to monitor the severity of depression and response to treatment.
Fear of cancer recurrence (FCR-1r) | Measured at baseline, 1-2 day(s) before surgery, perioperative (within 1 day of hospital discharge), 1, 3, 6 and 12 months post index surgery.
  Fear of cancer recurrence (FCR-1r) is a single-item screening measure for fear of cancer recurrence.The FCR-1r is a valid tool for FCR screening in colorectal cancer survivors with excellent ability to discriminate between clinical and non-clinical fear of cancer recurrence.
Adverse events (NHMRC Safety Monitoring and Reporting of Clinical Trials) | From date of opening recruitment to date of trial close-out
  The NHMRC publication Safety monitoring and reporting in clinical trials involving therapeutic goods sets out the requirements for the monitoring, collection and reporting of adverse events and adverse reactions that occur in clinical trials.
Self-efficacy (GSE) | Measured at 1, 3, 6 and 12 months post index surgery.
  General Self-Efficacy Scale (GSE) is a self-reported measure of self-efficacy.The General Self-Efficacy Scale is correlated to emotion, optimism, work satisfaction.The total score is calculated by finding the sum of the all items. For the GSE, the total score ranges between 10 and 40, with a higher score indicating more self-efficacy.
Treatment & Health Services | Measured at 1, 3, 6 and 12 months post index surgery.
  Data on treatments and health service utilisation including instance of treatment received, number of diagnostic imaging, number of GP/specialists visits, number of emergency department visits, number of hospital readmissions, number of support services received, hours of paid and unpaid work performed.
Satisfaction & Experience | Measured at 12 months post index surgery.
  Self-reported questionnaire asking participants to answer questions regarding their level of satisfaction with various components of the intervention reported on a 5-point Likert scale from extremely dissatisfied to extremely staisfied.
  Moreover, satisfaction feedback regarding the program, barriers and facilitators for future implementation will be obtained through interviews with clinicians, patients and caregivers at the end of the study period.
Return to work | Measured between 1 and 12 months post index surgery.
  Information about the impact of the intervention and surgery on return to work, and leisure activities will be obtained from questionnaires.
Acceptability of the intervention | Measured at 12 months post index surgery.
  Patients, clinicians and carers acceptability to the virtual multimodal hub (Intervention) will be assessed with a semi-structured questionnaire administered at 12-months (last survey). The semi-structured questionnaire contains 11 questions and participants (Patients, clinicians and carers) will be instructed to use a 5-point Likert Scale (ranked from strongly disagree to strongly agree) to express how much they agree or disagree with each statement. In addition, patients will be asked how satisfied they were with the virtual multimodal program and how confident they were in their ability to follow the advice given. The investigators will also take the opportunity to seek further feedback about the virtual multimodal hub (open ended question).

CONTACTS AND LOCATIONS:
Locations (31):
- Australia (31):
  - Coffs Harbour Health Campus, Coffs Harbour, New South Wales
  - Calvary Mater Hospital, Newcastle, New South Wales
  - John Hunter Hospital, Newcastle, New South Wales
  - Chris O'Brien Lifehouse, Sydney, New South Wales
  - Royal Prince Alfred Hospital, Sydney, New South Wales
  - Concord Repatriation General Hospital, Sydney, New South Wales
  - Westmead Hospital, Sydney, New South Wales
  - Blacktown Hospital, Sydney, New South Wales
  - Wagga Wagga Base Hospital, Wagga Wagga, New South Wales
  - Wollongong Hospital, Wollongong, New South Wales
  - Royal Brisbane & Women's Hospital, Brisbane, Queensland
  - Princess Alexandra Hospital, Brisbane, Queensland
  - The Queen Elizabeth II Jubilee Hospital, Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Flinders Medical Centre, Adelaide, South Australia
  - Modbury Hospital, Adelaide, South Australia
  - Lyell McEwin Hospital, Adelaide, South Australia
  - Grampians Health Ballarat Hospital, Ballarat, Victoria
  - Bendigo Health, Bendigo, Victoria
  - University Hospital Geelong (Barwon Health), Geelong, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Alfred Hospital, Melbourne, Victoria
  - Footscray Hospital, Melbourne, Victoria
  - Werribee Mercy Hospital, Melbourne, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria
  - St Vincent's Melbourne Hospital, Melbourne, Victoria
  - Northern Hospital Epping, Melbourne, Victoria
  - Austin Hospital, Melbourne, Victoria
  - Eastern (Box Hill) Hospital, Melbourne, Victoria
  - Cabrini Hospital, Melbourne, Victoria
  - Royal Perth Hospital, Perth, Western Australia

IPD SHARING:
Plan to Share IPD: Yes
Following explicit informed consent from individual participants, any de-identified data will be shared for studies approved by both the Principal Investigator (A/Prof Daniel Steffens) and a NHRMC approved Human Research Ethics Committee (HREC).
Supporting Information: Study Protocol, SAP
Time Frame: Data will only be made available upon individual request following the completion of the project. It will be at the discretion of the Principal Investigator (A/Prof Daniel Steffens) when this has been achieved. Once available, data may be accessed for up to 15 years after the trial's closure, after which it will be destroyed in accordance with the protocol.
Access Criteria: Based on explicit consent from individual participants, de-identified individual patient data (IPD) will be made available to researchers who comply with all regulations stipulated by a NHMRC-approved Human Research Ethics Committee (HREC). Subject to the discretion of both the Principal Investigator and a NHMRC-approved HREC, data will be made available for any approved analyses.
  Researchers interested in accessing IPD must submit a request to the Principal Investigator, A/Prof Daniel Steffens (daniel.steffens@health.nsw.gov.au). Mechanisms for data sharing will be in line with the Research Data Management Plan and a transfer process stipulated by a NHRMC approved HREC.